CLINICAL TRIAL: NCT05823051
Title: Akdeniz University
Brief Title: The Effect of Video-Assisted Sudden Infant Death Syndrome Prevention Training Program and Counseling Practice on Mothers' Knowledge Level and Self-efficacy: Randomized Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dilara Aydin Tozlu (Other)
Responsible Party: Sponsor-Investigator, Dilara Aydin Tozlu, Research Assistant, Akdeniz University
Organization: Akdeniz University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AUDilaraAT
Record Dates: First submitted 2023-04-08; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Sudden Infant Death
Keywords: Sudden Infant Death Syndrome; Nursing; Parent Education; Educational Program; Prevention
MeSH Terms: conditions — Sudden Infant Death

STUDY DESIGN:
Intervention Model Description: The study was planned as a randomized controlled, parallel, double centered and double blind study.
Who Masked: Participant, Outcomes Assessor
Masking Description: As a randomization method, "simple randomization method" will be used to ensure an equal number of samples in the two groups and to prevent bias. In addition, during the data analysis phase, the database will be created by an academician independent of the researcher providing the training.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VASIDS-TP and Counseling Practice (Experimental): Video-Assisted Sudden Infant Death Syndrome Prevention Training Program (VASIDS-TP) and Counseling Practice
  Interventions: Other: VASIDS-TP and Counseling Practice
- Routine Care (No Intervention): The control group will receive routine care in the obstetric ward. A pre-test will be conducted using the Google Survey form. "Personal Information Form", "Sudden Infant Death Syndrome Knowledge Level Assessment Form" (Pre-Test) and "General Self-Efficacy Scale" will be completed at this stage.
  The mothers in the control group will receive the training included in clinical routine care. The mothers in this group will not receive any planned structured training by the researchers during the study. The mothers in the control group will be administered the "Sudden Infant Death Syndrome Knowledge Level Assessment Data Form" and the "General Self-Efficacy Scale" with the Google survey that will be sent to their phones 1 month after the pre-test application. After the completion of the study, the control group will receive the same intervention (VASIDS-TP) as the intervention group.

INTERVENTIONS:
Other: VASIDS-TP and Counseling Practice — VASIDS-TP will be implemented online as an individual training to the intervention group through the Microsoft Teams program, to be completed in 5 days-5 sessions in the time frames determined by the participants. The consultancy practice will start with a pre-test and participants will be assured that they can call the researcher 24/7, and the consultancy practice will be continued by phone call or messaging.
  Arms: VASIDS-TP and Counseling Practice

SUMMARY:
Sudden Infant Death Syndrome (SIDS) is one of the leading causes of infant mortality in the postneonatal period, but it can be prevented and its incidence can be reduced by creating a safe sleep environment with modifiable risk factors. It is known that parents, infant care providers and healthcare professionals do not have sufficient knowledge about SIDS and safe sleep, and especially mothers exhibit many risky behaviors in terms of SIDS, such as using the wrong sleeping positions while putting their babies to sleep. Therefore, it is of critical importance to inform and raise awareness of parents on the issues of SIDS and safe sleep, which remain important today, on the premise of promoting public health.

DETAILED DESCRIPTION:
Sudden Infant Death Syndrome (SIDS) is one of the leading causes of infant mortality in the postneonatal period, but it can be prevented and its incidence can be reduced by creating a safe sleep environment with modifiable risk factors. It is known that parents, infant care providers and health professionals do not have sufficient knowledge about SIDS and safe sleep, and especially mothers exhibit many risky behaviors in terms of SIDS, such as using the wrong sleeping positions while putting their babies to sleep. Therefore, it is of utmost importance to inform and raise awareness of parents on the issues of SIDS and safe sleep, which remain important today, on the premise of promoting public health. In addition, informing mothers about the risk factors to protect their babies from SIDS, encouraging them to create and maintain a safe sleep environment, and ensuring that they are pioneers in this regard are also of great importance in terms of sharing information with other infant care providers in their social life. SIDS occurs in the postpartum period and has high values in infant mortality rates. For this reason, it is predicted that awareness on this issue will be significantly increased by providing education to new mothers at the earliest period and that SIDS can be prevented significantly by providing safe sleep environments. At the same time, based on the effect of self-efficacy perceptions of new mothers on the care of the baby, it is thought that the training and counseling practice planned to be given to mothers about SIDS will have a positive effect on the self-efficacy perceptions of mothers. When the relevant literature was examined, it was found that there were not enough studies on this subject in our country.

The aim of this study was to evaluate the effect of video-assisted Sudden Infant Death Syndrome prevention training program and counseling on mothers' knowledge level and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* The one who has just given birth,
* With a healthy newborn baby,
* Speaks, understands and can read and write Turkish and has no barriers to communication,
* Able to use the internet, telephone and e-mail actively,
* Mothers who voluntarily agreed to participate in the study will be included.

Exclusion Criteria:

* Have not attended at least 3 sessions of the training program,
* Mothers who indicate that they want to leave the study while the research is ongoing will be excluded.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — women who have just given birth
Enrollment: 80 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Sudden Infant Death Syndrome Knowledge Level Assessment Form 1 | Before the training
  This form was developed by the researchers in line with the literature and consists of 33 items to measure the level of knowledge about SIDS.
Sudden Infant Death Syndrome Knowledge Level Assessment Form 2 | 1 month after the training
  This form was developed by the researchers in line with the literature and consists of 33 items to measure the level of knowledge about SIDS.
General Self-Efficacy Scale 1 | Before the training
  "General Self-Efficacy Scale" is a five-point Likert-type scale consisting of 17 items. The question "How well does it describe you?" has five options ranging from "not at all" to "very well". The total score of the scale ranges between 17-85, and the higher the score, the higher the self-efficacy belief.
General Self-Efficacy Scale 2 | 1 month after the training
  "General Self-Efficacy Scale" is a five-point Likert-type scale consisting of 17 items. The question "How well does it describe you?" has five options ranging from "not at all" to "very well". The total score of the scale ranges between 17-85, and the higher the score, the higher the self-efficacy belief.

SECONDARY OUTCOMES:
Personal Information Form | Before the training
  The "Personal Information Form" developed by the researchers in line with the literature includes multiple-choice questions about mother, baby and sleep environment.
DISCERN Scale | After the training videos are created
  The training videos developed by the researchers will be evaluated by experts using DISCERN. Basically, it was developed to assess the quality of written and technology-based educational materials prepared to inform individuals about health and treatment options. The DISCERN scale consists of 16 items and each question is scored from 1 to 5. A score in the range of 15-75 is obtained by summing the responses from each item. In the evaluation, a low total score indicates poor quality and a high score indicates good quality.
System Usability Scale (SUS) | Pre-application
  In the test phase of the developed VASIDS-TP, SUS will be applied to evaluate the experiences of mothers (users). The whole scale consists of 10 questions. Each question has a value from 1 to 5 according to the answer given. SUS Score value is obtained between 0-100. SUS Score values of 68 points and above are considered above average, while values below 68 points are considered below average.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hutton JS, Gupta R, Gruber R, Berndsen J, DeWitt T, Ollberding NJ, Van Ginkel JB, Ammerman RT. Randomized Trial of a Children's Book Versus Brochures for Safe Sleep Knowledge and Adherence in a High-Risk Population. Acad Pediatr. 2017 Nov-Dec;17(8):879-886. doi: 10.1016/j.acap.2017.04.018. Epub 2017 Apr 24. PMID 28450082